CLINICAL TRIAL: NCT06374355
Title: Outcome of the Semibranch in Pararenal and Thoracoabdominal Aortic Pathologies. A Retrospective, Multicentre Registry
Brief Title: Semibranch Registry - Retrospective
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Alexander Oberhuber, Univ.-Prof. Dr. med., University Hospital Muenster
Other Study IDs: Semibranch_Retro
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Aortic Aneurysm; Endovascular Aortic Repair; Stent-Graft Endoleak
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Semibranch CMD branched aortic stentgraft — bEVAR with a custom made abdominal aortic multibranch, which incorporates the semibranch design

SUMMARY:
The goal of this registry is to evaluate the semibranch in branched endovascular arotic repair, which is a new tool in endovascular branched aortic repair.

DETAILED DESCRIPTION:
The main question it aims to answer are:

* Patency of the semibranch
* Feasibility of the technique regarding cannulation and stentgrafting

ELIGIBILITY:
* Patient has been treated with the semibranch stentgraft
* Patient is over 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pararenal or thoracoabdominal aortic pathology, who are treated with a endovascular semibranch stentgraft
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from target vessel instability | 30 days after intervention
  Primary patency and freedom from stenosis of the semibranch
Mortality | 30 days after intervention
  Overall mortality rate during 30 days after intervention
Technical success | 12 hours after intervention
  cannulation and stentgrafting ot the semibranches

SECONDARY OUTCOMES:
Morbidity | During follow up period (up to 3 years)
  Access site, bowel ischemia, kidney failure, paraplegia
Freedom of Endoleak type I and III | During follow up period (up to 3 years)
  Abscence of endoleaks arising from the semibranch
Long term mortality | During follow up period (up to 3 years)
  Overall mortality up to 3 years
Branch patency | During follow up period (up to 3 years)
  Primary patency of all branches

CONTACTS AND LOCATIONS:
Locations (1):
- Muenster University Hospital, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided